CLINICAL TRIAL: NCT02081066
Title: Relationship Between Endogenous CETP Activity and Atherosclerosis Distribution in Patients With High Cardiovascular Risk
Brief Title: Identification of CETP as a Marker of Atherosclerosis
Acronym: CETP-ATHERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C13-20; 2013-A00798-37 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-02-10; First posted 2014-03-07 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Heart Disease Risk Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with cardiovascular risk factors (Other)
  Interventions: Other: cardiovascular risk factors

INTERVENTIONS:
Other: cardiovascular risk factors

SUMMARY:
The reverse cholesterol transport (RCT) pathway, which involves the centripetal movement of free cholesterol from peripheral tissues, including the vessel wall, to the liver represent the primary mechanism by which HDL protects against atherosclerosis and by which it may induce plaque regression. Recent data reveal that the capacity of HDL to efflux cholesterol from macrophages, a metric of HDL function reflecting the initial step of the RCT, is clinically relevant, displaying a strong inverse association with both carotid intima-media thickness and the severity of angiographic CAD; such observations were independent of HDL-C levels.

In human, the Cholesteryl Ester Transfer Protein (CETP), represents a key protein of the RCT pathway and mediates redistribution of neutral lipids between lipoproteins, has been identified as a potential therapeutic target against atherosclerosis. It is known that CETP activity correlates with HDL-C levels and represents a key modulator of the ability of whole plasma to mediate free cholesterol efflux from human macrophages.

Recent studies showed that 23% of endogenous plasma CETP activity variability is explained by plasma LDL-C (12.0%), HDL-C (6.4%) and TG (4.4%) whereas sex and BMI accounted together for only 0.7% of its variability. Scoring patients for cardiovascular risk on the basis of their plasma lipid levels (TC, TG, LDL-C and HDL-C), revealed that patients with high cardiovascular risk (score ≥3) displayed a mean endogenous plasma CETP activity above 34%. Therefore plasma CETP activity represents a potent indicator of cardiovascular risk in patients with metabolic disorders since it integrates major independent risk factors.

The objective of this study is to decipher the relationship between CETP, HDL efflux capacity and the development of atherosclerosis in humans in order to identify CETP as a potent biomarker of atherosclerosis distribution.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of the study
* Men and women aged 18 or more years
* Patients displaying at least one abnormal plasma lipid parameter and/or receiving a lipid-lowering therapy unchanged for at least 3 months.

Exclusion Criteria:

* Current significant renal disease, including: nephrotic syndrome; chronic renal failure and/or serum creatinine >1.7 x upper limit of the reference range (ULRR)
* Uncontrolled hypothyroidism defined as TSH >2 x ULRR
* Active hepatobiliary disease, including chronic hepatitis B or hepatitis C infection (confirmed by serology); or an aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) >3.0 x ULRR
* Any prior history of malignancy or current cancer
* Current chronic or acute inflammatory syndrome defined as CRP>10 mg/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-09-25 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Endogenous CETP activity | Day 1
carotid intima-media thickness | day 1
Coronary calcium score | Day 1

SECONDARY OUTCOMES:
plasma efflux capacity from human macrophage | Day 1
HDL genetic variant | Day1

CONTACTS AND LOCATIONS:
Overall Officials: Maryse Guerin, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Inserm Umrs1166, Paris, France